CLINICAL TRIAL: NCT01192763
Title: A Neoadjuvant Pharmacodynamic Study Of RO4929097 (RO) in Pancreas Cancer
Brief Title: RO4929097 Before Surgery in Treating Patients With Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02523; NCI-2011-02523 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000683470; 10-089-A (Other: University of Chicago Comprehensive Cancer Center); 8522 (Other: CTEP); U01CA062505 (NIH); N01CM00071 (NIH)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Adenocarcinoma of the Pancreas; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Neoadjuvant Therapy

ARMS (1):
- Arm I (Experimental): Patients receive oral gamma-secretase inhibitor RO4929097 on days 1-3 and 8-10 in the absence of disease progression or unacceptable toxicity. Beginning 7 days after completion of gamma-secretase inhibitor RO4929097, patients undergo complete resection comprising pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy based on the anatomic location of the cancer. Tumor tissue from biopsy and surgery and blood samples are collected periodically for pharmacodynamic studies.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
This phase I trial is studying the side effects of RO4929097 before surgery in treating patients with pancreatic cancer. RO4929097 may stop the growth of tumor cells by blocking some enzymes needed for cell growth. Giving RO4929097 before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effects of neoadjuvant gamma-secretase inhibitor RO4929097 on Notch inhibition via interrogation of Hes-1 expression in patients with pancreatic cancer.

SECONDARY OBJECTIVES:

I. To evaluate the effects of this regimen on pancreatic cancer stem cell self-renewal and tumorigenesis as compared to pancreatic stem cells from controls (patients who do not receive treatment).

II. To evaluate the safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral gamma-secretase inhibitor RO4929097 on days 1-3 and 8-10 in the absence of disease progression or unacceptable toxicity. Beginning 7 days after completion of gamma-secretase inhibitor RO4929097, patients undergo complete resection comprising pancreaticoduodenectomy, distal pancreatectomy, or total pancreatectomy based on the anatomic location of the cancer. Tumor tissue from biopsy and surgery and blood samples are collected periodically for pharmacodynamic studies.

After completion of study therapy, patients are followed up every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * T1-3, N0-1, and M0 disease
* Surgically resectable disease confirmed by a surgeon experienced in pancreatic surgery

  * No borderline resectable disease defined as any of the following:

    * Tumors with severe unilateral or bilateral SMV/portal involvement impingement
    * Abutment (or) encasement of hepatic artery
    * SMA or celiac encasement (or) presence of SMV occlusion by tumor
* No metastatic disease
* ECOG performance status 0-1
* Life expectancy > 6 months
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 2 mg/dL
* Calcium, magnesium, phosphorous, and potassium normal
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective barrier-method contraception 4 weeks before, during, and for ≥ 12 months after completion of treatment
* Able to swallow tablets
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 or other agents used in the study
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia despite adequate electrolyte supplementation

  * Grade 1 hyponatremia with sodium ≤ 131 mg/dL is permissible
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia other than chronic
  * Stable atrial fibrillation
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Patients with a prior cancer with evidence of active cancer are excluded from this study

  * Patients with a prior cancer are permitted to enter this study as long as there is no documented evidence of active malignancy
* No uncontrolled electrolyte abnormalities including hypocalcemia, hypomagnesemia, and hypokalemia
* No symptomatic congestive heart failure, unstable angina pectoris, and a history of torsades de pointes or other significant cardiac arrhythmias
* No requirement for antiarrhythmics or other medications known to prolong QTc
* No other concurrent anticancer agents or therapies
* Recovered to < grade 2 toxicity related to prior therapy
* No prior chemotherapy or radiotherapy for pancreatic cancer
* No other concurrent investigational agents
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®), ketoconazole, or grapefruit juice
* No concurrent strong inducers or inhibitors of CYP3A4
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Notch activity (expression of Hes-1) | Up to day 3 (of course 1)
  Summarized as a binary endpoint for both the RO4929097 population and the stage-matched controls by the proportion and 95% exact binomial confidence interval.
Frequency and severity of adverse events as measured by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) | Up to 1 year
  Toxicity will be determined with a 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Proportion of cancer stem cells (CD44+, CD24+, ESA+ population of cells) self-renewal and tumorigenesis as measured by FACS | Up to day 3 (of course 1)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kim, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (6):
- United States (6):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Medical Center, Duarte, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - State Boulevard, Fort Wayne, Indiana